CLINICAL TRIAL: NCT04688632
Title: A Phase 1, Randomized, Double-Blind, Placebo- and Positive-Controlled, Thorough QT Study to Evaluate the Effect of Ampreloxetine on Cardiac Repolarization in Healthy Subjects
Brief Title: Thorough QT Study to Evaluate Ampreloxetine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0181
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypertension; nOH
Keywords: Symptomatic neurogenic orthostatic hypertension; nOH; Thorough QT; Symptomatic nOH
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1a (Active Comparator): Day 1: Single dose of Moxifloxacin Placebo; Day 1 - Day 15: Single daily dose of Ampreloxetine Placebo; Day 15: Single dose of Moxifloxacin <Dose A>
  Interventions: Drug: Ampreloxetine Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo
- Group 1b (Active Comparator): Day 1: Single dose of Moxifloxacin <Dose A>; Day 1 - Day 15: Single daily dose of Ampreloxetine Placebo; Day 15: Single dose of Moxifloxacin Placebo
  Interventions: Drug: Ampreloxetine Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo
- Group 2 - Treatment (Experimental): Day 1: Single dose of Moxifloxacin Placebo; Day 1 - Day 7: Single daily dose of Ampreloxetine <Dose A>; Day 8 - Day 14: Single daily dose of Ampreloxetine <Dose B>; Day 15: Single dose of Moxifloxacin Placebo; Day 15: Single dose of Ampreloxetine Placebo;
  Interventions: Drug: Ampreloxetine <Dose A>; Drug: Ampreloxetine <Dose B>; Drug: Ampreloxetine Placebo; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Ampreloxetine <Dose A> — Ampreloxetine <Dose A> will be administered as 1 tablet of <Dose A> and 3 tablets of Ampreloxetine Placebo.
  Arms: Group 2 - Treatment
Drug: Ampreloxetine <Dose B> — Ampreloxetine <Dose B> will be administered as 4 tablets of <Dose A>
  Arms: Group 2 - Treatment
Drug: Ampreloxetine Placebo — Ampreloxetine Placebo will be administered as 4 tablets of placebo. The placebo tablet will match (in appearance) the ampreloxetine <Dose A> tablet.
Drug: Moxifloxacin — Moxifloxacin will be administered orally as a single tablet.
  Arms: Group 1a; Group 1b
Drug: Moxifloxacin Placebo — Moxifloxacin placebo will be administered orally as a single tablet. The placebo tablet will match (in appearance) the moxifloxacin tablet.

SUMMARY:
A double-blind study to characterize the effect of ampreloxetine on cardiac repolarization in healthy subjects.

DETAILED DESCRIPTION:
A single-center, randomized, double-blind, placebo controlled, positive controlled, multiple dose, parallel group study will be conducted in healthy male and female subjects. Subjects will be randomized to one of 3 groups:

Subjects in Group 1a (n=18) will be administered moxifloxacin placebo on Day 1, ampreloxetine placebo from Day 1 to Day 15, and moxifloxacin <Dose A> on Day 15.

Subjects in Group 1b (n=18) will be administered a single oral dose of moxifloxacin <Dose A> on Day 1, ampreloxetine placebo from Day 1 to Day 15 and moxifloxacin placebo on Day 15.

Subjects in Group 2 (n=36) will be administered moxifloxacin placebo on Day 1 and on Day 15, and ampreloxetine <Dose A> from Day 1 to Day 7, ampreloxetine <Dose B> from Day 8 to Day 14, and ampreloxetine placebo on Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to give written informed consent.
2. Subject is a healthy, nonsmoking man or woman, 18 to 55 years of age, at screening.
3. Subject must be willing to abide by the following pregnancy precautions:

   * Female subjects must be either of non-childbearing potential or if of childbearing potential use a highly effective birth control method during the study and through 30 days after the last dose of study medication.
   * Male subjects (with partners of childbearing potential) must use acceptable contraception during the study and through 30 days after the last dose of study medication.
   * Subjects must agree not to donate ova or sperm during the study and for 30 days after the last dose of study medication.
4. Subject has a BMI of 18.0 to 30.0 kg/m2, inclusive, and weight of at least 55 kg at screening.
5. Subject has normal blood pressure (BP) and HR, measured after resting seated or supine for approximately 5 minutes. Normal BP is defined as 90 to 140 mmHg systolic and 50 to 90 mmHg diastolic. Normal HR is defined as 45 to 99 beats per minute (bpm) at screening and Day -2.
6. Subject is able to communicate well with the investigator and to comply with the study procedures, requirements, and restrictions.

Exclusion Criteria:

1. Subject has any clinically relevant abnormalities, as determined by the investigator, in the laboratory results at screening or Day -2. Except for the following clinical laboratory assessments outside the range specified:

   * hemoglobin <13.0 g/dL (men) or <11.5 g/dL (women),
   * hematocrit <38% (men) or <32% (women),
   * potassium <3.5 mEq/L,
   * magnesium <1.9 mg/dL, or
   * calcium <8.5 mg/dL
2. Positive results at screening for human immunodeficiency virus (HIV), hepatitis A virus (HAV) antibodies (anti-HAV: both IgG and IgM positive, IgG positive in the absence of IgM positive is acceptable), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody.
3. Within 4 weeks of screening and through Day 1, subject has:

   1. Confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (COVID-19) (test RT-PCR positive), OR
   2. Suspected SARS-CoV-2 infection (clinical features without documented test results) unless has a negative RT-PCR test for SARS-CoV-2 at least two weeks after resolution of symptoms and remains asymptomatic until Day 1, OR
   3. Close contact with a person with known or suspected SARS-CoV-2 infection unless has a negative RT-PCR test for SARS-CoV-2 at least two weeks after contact and remains asymptomatic until Day 1.
4. Subject has a prior history of myocardial infarction, acute coronary syndrome, cerebrovascular accident, transient ischemic attack, ventricular tachycardia, atrial fibrillation, personal or known family history of congenital long QT syndrome or known family history of sudden death with unknown cause prior to the age of 50, a pacemaker or implantable cardioverter defibrillator, cardiac or cerebral stent placement or angioplasty, or clinically significant valvular heart disease.
5. Subject has a history of orthostatic hypotension or orthostatic tachycardia or a history of dizziness, lightheadedness or fainting, or a feeling of blacking out upon standing, secondary to autonomic failure or other chronic cardiovascular condition.
6. Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematologic, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
7. Subject has a history of hypersensitivity to drugs (including moxifloxacin, related compounds, or excipients) with a clinically significant reaction or any clinically significant hypersensitivities.
8. Subject has any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract, including removal of parts of the stomach, bowel, liver, gall bladder [including cholecystectomy], or pancreas, but excluding procedures such as appendectomy and hernia repair).
9. Subject has participated in another clinical study of an investigational drug or medical device within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to screening, or is currently participating in another study of an investigational drug or medical device.
10. Subject is unwilling to abstain from ingestion of caffeine or xanthine-containing products (e.g., tea, coffee, chocolate, cola, etc.) beginning 48 hours prior to admission to the CRU on Day -2 until the final PK sample has been collected.
11. Subject is unwilling to abstain from alcohol beginning 48 hours prior to admission to the CRU on Day -2 until the final PK sample has been collected.
12. Subject has a history of drug abuse (in the past 3 years) or positive screen for drugs of abuse or alcohol at screening or on Day -2.
13. Subject has a history of alcohol consumption within 6 months prior to screening, defined as an average weekly intake of >14 units for males or >10 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine, or 1 measure (25 mL) of spirits.
14. Subject uses or has used tobacco-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) within 6 months prior to screening or has a positive cotinine result at screening or on Day -2 and is unwilling to abstain from tobacco containing products until follow-up.
15. Subject has consumed grapefruit (or Seville Oranges) and/or grapefruit juice or food containing grapefruit (or Seville oranges [e.g., orange marmalade]), within 14 days prior to admission to the CRU on Day -2 and is unwilling to abstain from consuming these items until the final PK sample has been collected.
16. Subject has consumed other fruit juices within 48 hours prior to admission to the CRU on Day -2 and is unwilling to abstain from these items until the final PK sample has been collected.
17. Subject has consumed cruciferous vegetables (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard greens) or charbroiled meats within 7 days prior to admission to the CRU on Day -2 and is unwilling to abstain from these items until the final PK sample has been collected.
18. Subject is unwilling to abstain from any strenuous physical exercise (such as weight training, aerobics) 24 hours prior to admission to the CRU on Day -2 until the final PK sample has been collected.
19. Subject has acute illness (gastrointestinal illness, infection [e.g., influenza] or known inflammatory process) at screening or within 2 weeks prior to admission to the CRU on Day 2.
20. Subject uses any prescription drug or over-the-counter medication, including herbals or routine vitamins or minerals within 14 days or 5 half-lives (whichever is longer) prior to admission to the CRU on Day -2 or subject requires continued use of a prescription drug or over-the-counter medication during study participation.
21. Subject has donated blood or had blood loss of more than 400 mL or blood components within the 8 weeks prior to screening or plans to donate blood during the study.
22. Subject has a clinically significant abnormal screening ECG indicating a second- or third degree atrioventricular block, or one or more of the following: QRS >110 msec, QT interval corrected using Fridericia's formula (QTcF) >440 msec (men and women), PR interval >200 msec.
23. Subject has any significant morphological changes other than minor nonspecific T wave changes in the opinion of the investigator, including flat T waves in the inferior leads, which are interpreted by the investigator to interfere with QT analysis or to be clinically significant.
24. Subject has a known hypersensitivity towards medications similar to ampreloxetine or excipients contained in ampreloxetine.
25. Subject has previously participated in a study for ampreloxetine.
26. Subject has demonstrated a history of lifetime suicidal ideation and/or suicidal behavior, as outlined by the C-SSRS (Baseline/Screening Version) subject should be assessed by the rater for risk of suicide and the subject's appropriateness for inclusion in the study.
27. Subject, who, for any reason, is deemed by the investigator to be inappropriate for this study or has any condition which would confound or interfere with the evaluation of the safety, tolerability, or pharmacokinetics of the investigational drug or prevent compliance with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
QTcF | Days -1, 1, 7, 8, 14 and 15
  Change in QTcF from baseline

SECONDARY OUTCOMES:
Cmax | Day 1 to Day 16
  Maximum observed plasma concentration (Cmax) for ampreloxetine
Tmax | Day 1 to Day 16
  Time to reach maximum observed plasma concentration (Tmax) for ampreloxetine
AUC0-24 | Day 1 to Day 16
  Area under the concentration time curve during 0-24 hours (AUC0-24) for ampreloxetine
ECG - HR | Days -1, 1, 7, 8, 14 and 15
  Change-from-baseline in Electrocardiogram (ECG) - Heart Rate (HR)
ECG - PR Interval | Days -1, 1, 7, 8, 14 and 15
  Change-from-baseline in Electrocardiogram (ECG) - PR Interval
ECG - QRS Interval | Days -1, 1, 7, 8, 14 and 15
  Change-from-baseline in Electrocardiogram (ECG) - QRS Interval

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.